CLINICAL TRIAL: NCT03697460
Title: INCB018424 in the Treatment of Cutaneous Lichen Planus
Brief Title: Topical Ruxolitinib Lichen Planus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aaron R. Mangold (Other)
Responsible Party: Sponsor-Investigator, Aaron R. Mangold, Assistant Professor of Dermatology, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-005406
Record Dates: First submitted 2018-10-03; First posted 2018-10-05 (Actual); Results first posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Lichen Planus
MeSH Terms: conditions — Lichen Planus | interventions — ruxolitinib

STUDY DESIGN:
Intervention Model Description: Topical INCB018424
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INCB018424 (Experimental): INCB018424 Cream
  Interventions: Drug: INCB018424

INTERVENTIONS:
Drug: INCB018424 — INCB018424 PHOSPHATE CREAM 1.5%, topical application, twice daily on lesions of cutaneous LP.

SUMMARY:
To evaluate the safety and efficacy of INCB018424 PHOSPHATE CREAM in cutaneous LP as assessed by the change in Physician Global Assessment (PGA), Body Surface Area (BSA), Index Treatment and Control Lesion by Clinical Assessment Scale of Severity for Index Lesion Signs and Symptoms (CAILS) score, Pruritus Numerical Rating Scale (NRS), and Skindex-16. To predict responses through the identification of unique biomarkers of LP at week 0 and utilizing RNA sequencing on responsive and non-responsive tissue at week 4.

DETAILED DESCRIPTION:
This is a single center, exploratory, open-label, single-arm design study of 12 patients. Treatment naïve and treatment refractory patients with LP will be treated with INCB018424 PHOSPHATE CREAM. Patients who are non-responders, to physician choice standard of care, will undergo a washout period and will be enrolled in the study. The study consists of 3 epochs: screening/washout period (of at least 1 week and up to 4 weeks), treatment epoch (of 8 weeks from screen/washout), and follow up epoch (of 4 weeks). The screening and washout period will allow for treatment naïve/ new diagnosis LP to undergo evaluation and diagnosis and for treatment refractory to undergo a washout. The total duration of the study will be 13-16 weeks.

ELIGIBILITY:
Subjects must be able to understand and comply with the requirements of the study and communicate with the investigator.

Subjects must give written, signed, and dated informed consent before any study related activity is performed.

When appropriate, a legal representative will sign the informed consent according to local laws and regulation

Both men and women must be at least 18 years of age at the time of screening

Subjects must have clinical and histological features of LP

LP must involve between 2 and 20% of the BSA

Subjects must have a minimum of 10 lesions of LP

Subjects must have treatment naive cutaneous LP or treatment refractory disease, as defined by failure of at least one established treatment for LP

Failure of prior therapy Topical treatment Systemic immunosuppressant Oral metronidazole Oral sulfasalazine Oral retinoid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron R Mangold, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brumfiel CM, Patel MH, Severson KJ, Zhang N, Li X, Quillen JK, Zunich SM, Branch EL, Nelson SA, Pittelkow MR, Mangold AR. Ruxolitinib Cream in the Treatment of Cutaneous Lichen Planus: A Prospective, Open-Label Study. J Invest Dermatol. 2022 Aug;142(8):2109-2116.e4. doi: 10.1016/j.jid.2022.01.015. Epub 2022 Feb 5. PMID 35131254
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- INCB018424: Subjects applied INCB018424 topically, twice daily.
  INCB018424 Cream
  INCB018424: INCB018424 PHOSPHATE CREAM 1.5%, topical application, twice daily on lesions of cutaneous LP.
Period: Overall Study
Arm/Group | INCB018424
Started | 12
Completed | 9
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | INCB018424
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 63 [34 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 11
  Hispanic | 1
Region of Enrollment [Number; unit: participants]
  United States | 12
Duration of Disease [Mean (Standard Deviation); unit: years] | 1.25 (1.13)
Number of Prior Treatments [Mean (Standard Deviation); unit: prior treatments] | 2.2 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Modified Clinical Assessment Scale of Severity for Index Lesion Signs and Symptoms (mCAILS)
Description: mCAILS summation score as measured by Erythema (0-8), Scaling (0-8) Plaque elevation (0-8) Hyper/hypopigmentation (0-8) Size (0-18), Total score ranging from 0-50 with higher score indicating higher severity
Time Frame: week 0, week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | INCB018424
Number analyzed (Participants) | 12
score on a scale | 11.0 (6.2)

2. Primary Outcome: Change in Total Body Lesion Count
Description: The number of total body lesions.
Time Frame: week 0, week 4
Measure: Median (Inter-Quartile Range); unit: lesions
Arm/Group | INCB018424
Number analyzed (Participants) | 12
lesions | 50 [25 to 723]

3. Secondary Outcome: Change in Pruritus Numerical Rating Scale
Description: Pruritus Numerical Rating Scale as measured by they question "How severe has your itching been over the last 24 hours?" Ranging from 0 = none, to 10 = severe. The higher the score the more severe.
Time Frame: week 0, week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | INCB018424
Number analyzed (Participants) | 12
score on a scale | 4.4 (3.0)

4. Secondary Outcome: Change in Overall Quality of Life Skindex-16 Score
Description: Skindex-16 score as measured by 16 questions, 3 subscales: Symptoms, Emotional, Functional. Score ranges for each question (0-6). Total score ranging from 0-96 with higher score indicating worse quality of life
Time Frame: week 0, week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | INCB018424
Number analyzed (Participants) | 12
score on a scale | 36.3 (17.5)

5. Secondary Outcome: Number of Subjects With Greater Than or Equal to 50% Improvement in Physician Global Assessment Score
Description: PGA score as measured by Grade 0 (clear: no evidence of disease (100% improvement)) to Grade 6 (Worse, disease is worse than at baseline evaluation by (≥25%) or more). Higher score equals worse disease
Time Frame: week 0, week 4
Measure: Number; unit: participants
Arm/Group | INCB018424
Number analyzed (Participants) | 12
participants | 12

6. Secondary Outcome: Body Surface Area (BSA) Affected by Cutaneous Lichen Planus
Description: BSA as measured as the percentage of the body affected by Cutaneous Lichen Planus. Ranging from 0-100% of the body.
Time Frame: week 0, week 4
Measure: Mean (Standard Deviation); unit: mean percentage of body surface area
Arm/Group | INCB018424
Number analyzed (Participants) | 12
mean percentage of body surface area
  Week 0 | 6.1 (7.9)
  Week 4 | 0.9 (1.9)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 12 weeks.
Arm/Group | INCB018424
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 7/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INCB018424 (N=12)
Abnormal Taste (Nervous system disorders) | 1 (1)
Blood Clot (Blood and lymphatic system disorders) | 1 (1)
Cold (General disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Incontinence (Renal and urinary disorders) | 1 (1)
Light headedness (Nervous system disorders) | 1 (1)
Sleep Disturbance (Psychiatric disorders) | 1 (1)
Pressure on right arm (Musculoskeletal and connective tissue disorders) | 1 (1)
Sinus Infection (Infections and infestations) | 1 (1)
Vaginal Infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Yeast Infection (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
All subjects reached the 4 week endpoint. Due to surrounding the Covid-19 pandemic, 2 subjects did not complete weeks 8 or 12 and 1 subject did not complete week 12.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/60/NCT03697460/Prot_SAP_000.pdf